CLINICAL TRIAL: NCT03890419
Title: Opioid Sparing Potential of Light-Induced Analgesia: a Pilot Trial of a Novel, Non-Pharmacological Treatment for Pain
Brief Title: Opioid Sparing Potential of Light-Induced Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00102106
Record Dates: First submitted 2019-03-21; First posted 2019-03-26 (Actual); Results first posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Pain
Keywords: Acute Pain; Chronic Pain; Opioid Use; Pain
MeSH Terms: conditions — Pain; Acute Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Control Group participants will be exposed to full spectrum light during the study.
  Interventions: Device: Clear light
- Green light Group (Experimental): Green light Group participants will be exposed to green light during the study.
  Interventions: Device: Green light
- Blue light Group (Experimental): Blue light Group participants will be exposed to blue light during the study.
  Interventions: Device: Blue Light

INTERVENTIONS:
Device: Green light — Green light exposure
  Arms: Green light Group
Device: Clear light — Full spectrum light exposure
  Arms: Control Group
Device: Blue Light — Blue light exposure
  Arms: Blue light Group

SUMMARY:
This is a pilot trial testing the potential opioid-sparing analgesic effect of a novel non-pharmacological treatment using visualized light spectrums. Preclinical findings have shown such treatments to alter pain perception.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for thoracic surgery for which post-operative opioid PCA is anticipated (Acute Pain group) OR currently treated with opioid therapy for fibromyalgia (Chronic Pain group)
* 18 years of age and older
* Able to wear study eyeglasses for at least 4 hours per day
* Agree to participate and provide written informed consent and HIPAA authorization

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Padma Gulur, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health Systems, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Green Light Group | Blue Light Group
Started | 34 | 30 | 30
Completed | 27 | 27 | 25
Not Completed | 7 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Green Light Group | Blue Light Group | Total
Number analyzed (Participants) | 34 | 30 | 30 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 22 | 61
  >=65 years | 14 | 11 | 8 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (10.2) | 59.2 (13.8) | 53.9 (12.8) | 57.9 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 21 | 66
  Male | 12 | 7 | 9 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 32 | 30 | 29 | 91
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 10 | 7 | 8 | 25
  White | 23 | 18 | 20 | 61
  More than one race | 1 | 4 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 30 | 30 | 94

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Level
Description: Pain level assessed using the Numeric Rating Scale. In a Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10 that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'. Primary assessment is day 1 compared to end of study assessment (week 2 in chronic pain and 48 hours in acute pain). The end of study values were averaged with standard deviation for all patients at their end of study assessment.
Time Frame: Baseline to end of study
Population: Participants with available data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Green Light Group | Blue Light Group
Number analyzed (Participants) | 27 | 25 | 25
score on a scale | 1.15 (2.84) | -0.04 (1.88) | 1.07 (2.33)

2. Primary Outcome: Change in Opioid Dose Used for Pain
Description: Change in amount of opioid medication used for pain relief measured in oral morphine equivalents. Primary assessment is day 1 compared to end of study assessment (week 2 in chronic pain and 48 hours in acute pain). The end of study values were averaged with standard deviation for all patients at their end of study assessment.
Time Frame: Baseline to end of study
Population: Participants with available data.
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Control Group | Green Light Group | Blue Light Group
Number analyzed (Participants) | 27 | 25 | 25
MME | 37.36 (68.23) | 37.38 (76.03) | 56.20 (151.11)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from consent through follow-up study visit (2 weeks)
Arm/Group | Control Group | Green Light Group | Blue Light Group
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 6/34 | 0/30 | 2/30
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=34) | Green Light Group (N=30) | Blue Light Group (N=30)
Headache/Migraine (General disorders) | 6 (6) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT03890419/Prot_SAP_001.pdf
  • Informed Consent Form (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT03890419/ICF_000.pdf